CLINICAL TRIAL: NCT07080437
Title: An Observational Study on the Safety and Efficacy of Immunotherapy Combined With Concurrent Chemoradiotherapy in Elderly Patients With Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Three Gorges Hospital of Chongqing University (Other)
Responsible Party: Principal Investigator, HanZhang, Doctor, Three Gorges Hospital of Chongqing University
Other Study IDs: TGHEC001
Record Dates: First submitted 2025-07-08; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Immunotherapy Therapy — Patients will receive concurrent chemoradiotherapy (CCRT) combined with immunotherapy. The treatment includes:
  Radiotherapy: Individualized radiotherapy targeting the tumor. Concurrent Chemotherapy: Platinum-based doublet chemotherapy (e.g., cisplatin + fluorouracil or S-1) administered during radiotherapy.
  Immunotherapy: PD-1 inhibitor (e.g., tislelizumab) used to enhance the immune response against cancer cells.
  The treatment will be tailored to each patient's condition, with regular follow-up assessments every 3 months for up to 2 years to monitor efficacy and safety.

SUMMARY:
Title: Observational Study on the Safety and Efficacy of Immunotherapy Combined with Concurrent Chemoradiotherapy in Elderly Patients with Esophageal Squamous Cell Carcinoma

Study Purpose:

This single-center, open-label, retrospective study aims to evaluate the safety and efficacy of immunotherapy combined with concurrent chemoradiotherapy (CCRT) in elderly patients with esophageal squamous cell carcinoma (ESCC). The primary objectives include assessing the objective response rate (ORR), overall survival (OS), progression-free survival (PFS), disease control rate (DCR), duration of response (DoR), R0 resection rate, adverse events (AEs), and potential predictive biomarkers in elderly patients receiving this treatment regimen.

Condition Studied:

Esophageal Squamous Cell Carcinoma (ESCC) in elderly patients (≥70 years).

Intervention:

Participants will receive concurrent chemoradiotherapy (CCRT) combined with immunotherapy. The study will retrospectively analyze the outcomes of patients treated between January 2022 and March 2025.

Study Design:

This is a retrospective, single-arm study. Patients aged 70 years or older with histologically confirmed ESCC (stages IB to IVB according to the 6th edition of the American Joint Committee on Cancer) will be included. Patients will undergo radiotherapy with concurrent chemotherapy and immunotherapy. Follow-up evaluations will be conducted every 3 months until disease progression or up to 2 years.

Eligibility Criteria:

Inclusion Criteria:

Voluntary participation with written informed consent. Age ≥70 years, regardless of gender. Histologically or cytologically confirmed ESCC. Inoperable or refusal of surgery, with tolerance for anti-tumor treatment. ECOG performance status 0-2. Expected survival ≥6 months. No severe abnormalities in hematologic, cardiac, pulmonary, hepatic, or renal function, and no immunodeficiencies.

Exclusion Criteria:

Distant organ metastasis (excluding supraclavicular lymph nodes). Previous esophageal fistula, perforation, or pre-treatment for malignancy. Prior thoracic radiotherapy. Active autoimmune diseases or history of autoimmune diseases. Previous or ongoing PD-1 inhibitor treatment or participation in other interventional clinical studies.

Allergy to large protein formulations or components of S-1 capsules. Uncontrolled cardiac conditions. Immunodeficiencies (e.g., HIV infection), active hepatitis B or C, or active tuberculosis.

Active infection or unexplained fever >38.5°C within 2 weeks before screening. History of other malignancies within 5 years (except cured basal cell carcinoma of the skin or cervical carcinoma in situ).

Scientific and Social Value:

This study aims to explore effective treatment options for elderly ESCC patients and enhance the influence of the discipline in this field.

Recruitment and Informed Consent:

Participants will be recruited through physician referrals. Informed consent will be obtained from all participants, ensuring their privacy and confidentiality.

Outcome Measures:

Primary outcomes: ORR, OS, PFS, DCR, DoR, R0 resection rate, and AEs. Secondary outcomes: Identification of potential predictive biomarkers.

Study Duration:

The study will cover a period from January 2022 to March 2025, with follow-up evaluations conducted every 3 months until disease progression or up to 2 years.

Publication Plan:

The results of this study will be published in high-quality scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation with written informed consent. Age ≥70 years, regardless of gender. Histologically or cytologically confirmed ESCC. Inoperable or refusal of surgery, with tolerance for anti-tumor treatment. ECOG performance status 0-2. Expected survival ≥6 months. No severe abnormalities in hematologic, cardiac, pulmonary, hepatic, or renal function, and no immunodeficiencies.

Exclusion Criteria:

* No severe abnormalities in hematologic, cardiac, pulmonary, hepatic, or renal function, and no immunodeficiencies.

Exclusion Criteria:

Distant organ metastasis (excluding supraclavicular lymph nodes). Previous esophageal fistula, perforation, or pre-treatment for malignancy. Prior thoracic radiotherapy. Active autoimmune diseases or history of autoimmune diseases. Previous or ongoing PD-1 inhibitor treatment or participation in other interventional clinical studies.

Allergy to large protein formulations or components of S-1 capsules. Uncontrolled cardiac conditions. Immunodeficiencies (e.g., HIV infection), active hepatitis B or C, or active tuberculosis.

Active infection or unexplained fever >38.5°C within 2 weeks before screening. History of other malignancies within 5 years (except cured basal cell carcinoma of the skin or cervical carcinoma in situ).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of elderly patients (≥70 years) with histologically confirmed ESCC who are not suitable for surgery or refuse surgery but are able to tolerate anti-tumor treatment. The inclusion and exclusion criteria are designed to ensure the safety and efficacy of the study while maintaining a representative patient population for the research objectives.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 months
  Imaging assessments every 3 months after treatment initiation until disease progression or up to 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Shangxia Hospital of Chongqing University, Chongqing, Chongqing Municipality, China